CLINICAL TRIAL: NCT06830239
Title: Early Phase II Exploratory, Open-Label, Non-Randomized Study of Neoadjuvant Dostarlimab Monotherapy in Participants With Untreated T3-4N0-2 or Stage III pMMR/MSS Resectable Colon Cancer
Brief Title: Phase II Study of Neoadjuvant Dostarlimab in Patients With Untreated T3-4N0-2 or Stage III pMMR/MSS Resectable Colon Cancer
Acronym: Superhero
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S68882; 2024-512499-36-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-10; First posted 2025-02-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colon Cancer Stage III
Keywords: Colon Cancer; Neoadjuvant; pMMR/MSS; Resectable
MeSH Terms: conditions — Colonic Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dostarlimab monotherapy (Experimental): Dostarlimab should be administered by intravenous infusion using an intravenous infusion pump over 30 minutes at a dose of 500 mg once every 3 weeks (Q3W), for 2 cycles (6 weeks in total).
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — Dostarlimab [Jemperli GlaxoSmithKline (GSK)] is a humanized IgG4 monoclonal antibody that binds with high affinity and specificity to PD-1, resulting in inhibition of binding to PD-L1 and PD-L2.
  Dostarlimab is in clinical development for the treatment of subjects with solid tumors, including those with recurrent/advanced dMMR/MSI-H solid tumors who have progressed on standard of care chemotherapy, as monotherapy or in combination with other agents.
  Other Names: Jemperli

SUMMARY:
Dostarlimab belongs to a class of drugs called PD-1 inhibitors that use your own immune system to treat cancer (immunotherapy). It is designed to stop cancer from growing by helping your immune system recognize and fight the cancer. This investigational medicinal product (IMP) has been approved by the Belgian authorities, but not for the treatment of colon cancer.

It is known that a small number of patients with pMMR/MSS colon cancer may have significant response to medication of this type (immunotherapy) depending on each person's biology.

Trial intervention for all patients will be neo-adjuvant dostarlimab 500 mg IV, given alone by intravenous infusion. Two administrations of dostarlimab are foreseen, at three weeks interval, before surgery for your colon cancer. It has not yet been proven that this treatment can cure, improve or stabilise your disease or condition.

The study aims to investigate specific molecular changes in tumour and blood after dostarlimab monotherapy administered and before surgery which could be associated with improved response to conventional treatment in some patients. If you decide to participate, as the duration of treatment with dostarlimab is 6 weeks, surgery may be slightly delayed compared to patients that are not treated with dostarlimab and go directly for surgery. It remains uncertain if this is beneficial in your personal situation but some patients might experience significant response. The risks have been carefully assessed and the potential benefits for some patients are considered important and justify undertaking the treatment.

Subsequent therapy after surgery remains at the discretion of the treating physician.

The duration of a patient on trial will last up to 4 months from the first dose of dostarlimab and afterwards 2 years of follow up is applicable.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age and capable of giving informed consent
* primary adenocarcinoma colon cancer than can be removed surgically, staged cT3-4, cN0-2, cM0 or stage III
* tumour expresses an MMR proficient/microsatellite stable called MSS
* tissue samples from tumour and colon mucosa available for molecular analyses
* capable of receiving immunotherapy
* adequate general health status and organ function (blood tests)

Exclusion Criteria:

* no prior cancer treatment
* not pregnant and using effective contraception if applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Multi-omic exploration | From enrollment to the last FU visit of the patient for blood (2 years). From baseline to surgery for tissue (12-15 weeks). Data will be reported at the final study report (max 3 years from study start).
  Data generation through multi-omic exploration of blood and tissue derived products (see Sampling and Lab manual). Correlation of molecular-biological features identified with pathological response. The presence or absence of specific molecular characteristics in blood and tissue will be correlated in each patient with the degree of tumour response to therapy evaluated by a pathologist.

SECONDARY OUTCOMES:
Safety analysis | Continuous
  Safety analysis. Frequency and severity of treatment emergent AEs, SAEs, irAEs. AEs leading to death, discontinuation of trial intervention or resulting in the participant not being suitable for surgery.
Pathological response | Pathological tumor staging and response assessment is at surgery
  Proportion of participants with pathological response, determined by local assessment.
Survival | From enrollment till last FU visit of patient (2 years). Data will be reported at the final study report (max 3 years from study start).
  Survival time defined from Superhero ICF signature to death from any cause. Proportion of survivors at 2 years.
  Event free survival time (EFS) defined from Superhero ICF signature to recurrence evaluated by local assessment or death.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Tejpar, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided